CLINICAL TRIAL: NCT01311232
Title: Hepatitis B Virus Reactivation in Asian Patients Treated With Rituximab-containing Treatment
Brief Title: Factors Influencing Hepatitis B Virus Reactivation in Lymphoma Patients Treated With Rituximab
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, Professor, Samsung Medical Center
Other Study IDs: 2010-11-035
Record Dates: First submitted 2011-03-06; First posted 2011-03-09 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Patients With Diffuse Large B-cell Lymphoma or Follicular Lymphoma; Patients Treated With Rituximab-CHOP or Rituximab-CVP
Keywords: rituximab, lymphoma, hepatitis B virus
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma; Hepatitis B

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Case: Patients with HBV reactivation
- Control: Patients without HBV reactivation

SUMMARY:
This study is a retrospective analysis to identify factors influencing hepatitis B virus reactivation in patients treated with rituximab containing chemotherapy. Rituximab monoclonal antibody targeting CD20 induces B-cell depletion resulting in prolonged immune suppression. This leads to frequent reactivation of patients with a previous history of exposure to HBV or HBV carrier.

We collect the clinical features and laboratory findings of patients satisfied the inclusion criteria as follows.

1. Patients diagnosed with diffuse large B-cell lymphoma (DLBCL) or \ follicular B-cell lymphoma (FL).
2. Patients who had received at least two cycles of rituximab-CHOP or rituximab-CVP as a primary treatment
3. Patients with a history of previous exposure to HBV

   * HBV surface antigen (HBs Ag) positive Or
   * HBV core antibody (IgG anti-HBc antibody) positive

Then, we compare the HBV reactivation group with the control group (HBV reactivation does not happen) to find factors influencing HBV reactivation.

DETAILED DESCRIPTION:
Description of factors associated with Hepatitis B virus reactivation:

* Laboratory parameters defining HBV status/activity at time of treatment initiation
* Lymphoma stage at rituximab treatment initiation (Ann Arbor, B-symptoms, bone marrow involvement, IPI, ECOG-score, LDH)
* Immunochemotherapy regimen (treatment line, rituximab dose and cycle)
* Disease status at time of HBV reactivation
* Antiviral prophylaxis (medication, dose, duration at time at time of reactivation)
* Patient demographics (age, gender, residence, ethnic origin, smoking status, alcohol consumption and occupation)

Time to Hepatitis B virus reactivation

* The time from start of rituximab-containing immunochemotherapy until first evidence of HBV reactivation meeting the criteria
* Description of prophylaxis and treatment with antiviral medication HBV vaccination Time of initiation of antiviral therapy of prophylaxis relating to clinical or laboratory signs of possible HBV reactivation Anti-viral medication used in prophylaxis or therapy
* Description of outcomes Outcomes of the HBV reactivation Outcomes of the rituximab-containing immunochemotherapy Demographics and previous infection history: Age, gender, nationality, race, social history, past medical history
* Parameters associated with lymphomas: Ann Arbor stage, number of extranodal involvement, serum LDH, serum β2-microglobulin, ECOG performance status, presence of B symptoms, International Prognostic Index, bone marrow invasion
* Laboratory parameters associated with hepatitis B virus:

hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (anti- HBs), hepatitis B e antigen (HBeAg), hepatitis B core antibody (anti-HBc), hepatitis B e antibody (anti-HBe), serum HBV DNA

* Lymphoma treatment history:

Line of treatment (first line, second line), rituximab and chemotherapy administration (dose, schedule), start date, last treatment date

* Prophylaxis or treatment against HBV reactivation:

antiviral drug (dose, schedule, duration)

* Hepatitis B virus reactivation:

onset, serologic markers, outcome

ELIGIBILITY:
Inclusion Criteria

1. Patients diagnosed with diffuse large B-cell lymphoma (DLBCL) or follicular B-cell lymphoma (FL).
2. Patients who had received at least two cycles of rituximab-CHOP or rituximab-CVP as a primary treatment
3. Patients with a history of previous exposure to HBV

   * HBV surface antigen (HBs Ag) positive Or
   * HBV core antibody (IgG anti-HBc antibody) positive
4. Patients with documented HBV reactivation (definite or presumptive) occurring during treatment (at least two cycles of R-CHOP or R-CVP) or within 12 months after the last dose of rituximab

   * Definitive HBV reactivation

     - Elevation of serum HBV DNA level >1 log IU/mL from baseline or absolute increase of HBV DNA by 6 log10 IU/mL in HBsAg positive patients
   * Presumptive HBV reactivation - Increase of ALT (≥3x baseline value or absolute value of ≥100 U/L) and positive conversion of HBs Ag in previously HBsAg-negative patients

Exclusion Criteria:

1. Patients who had received chemotherapy other than R-CHOP or R-CVP after diagnosis
2. patients diagnosed with HIV, HCV or HDV co-infection
3. Patients who had undergone allogenic stem cell transplantation before hepatitis B virus reactivation was documented

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hepatitis B virus positivity and treated with rituximab-containing chemotherapy to treat their disease, diffuse large B-cell lymphoma or follicular lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2010-11-01 (Actual); Primary Completion 2012-12-01 (Actual); Study Completion 2013-12-01 (Actual)

PRIMARY OUTCOMES:
Hepatitis B virus reactivation | one year

CONTACTS AND LOCATIONS:
Locations (4):
- Queen Mary Hospital, Hing Kong, China
- Hospital Kuala Lumpur, Kuala Lumpur, Malaysia
- National Cancer Center, Singapore, Singapore
- Samsung Medical Center, Seoul, South Korea